CLINICAL TRIAL: NCT07181109
Title: ZENITH: A Phase 3 Global, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Zilebesiran in Addition to Standard of Care in Reducing Major Adverse Cardiovascular Events in Adult Patients With Hypertension Not Adequately Controlled and With Either Established Cardiovascular Disease or High Risk for Cardiovascular Disease
Brief Title: Zilebesiran in Patients With Hypertension Not Adequately Controlled and With Either Established Cardiovascular Disease or High Risk for Cardiovascular Disease
Acronym: ZENITH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-AGT01-008; 2025-522960-34-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: High Risk Cardiovascular Disease; Hypertension; High Cardiovascular Risk
Keywords: High blood pressure; siRNA; Angiotensinogen; AGT; Cardiovascular disease; Uncontrolled hypertension; RNAi
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zilebesiran 300 mg (Experimental): Participants will be administered 300 mg zilebesiran subcutaneously (SC) once every 6 months as add-on therapy to their standard of care antihypertensive medications.
  Interventions: Drug: Zilebesiran
- Placebo (Placebo Comparator): Participants will be administered placebo SC once every 6 months as add-on therapy to their standard of care antihypertensive medications.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zilebesiran — Zilebesiran will be administered SC
  Other Names: ALN-AGT01
  Arms: Zilebesiran 300 mg
Drug: Placebo — Placebo will be administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether zilebesiran versus placebo reduces the risk of cardiovascular (CV) death, nonfatal myocardial infarction (MI), nonfatal stroke, or heart failure (HF) events. This is an event-driven study that will continue until the targeted number of positively adjudicated primary endpoint clinical outcome events (COEs) have been reached.

ELIGIBILITY:
Inclusion Criteria:

* Is 18 years or older for patients with established cardiovascular disease (CVD)
* Is 55 years or older for patients with high risk for CVD
* Has established CVD (defined as coronary, cerebrovascular, or peripheral artery disease) or high risk for CVD
* Has treated hypertension on stable therapy with at least 2 standard of care antihypertensive medications, one of which must be a thiazide, thiazide-like, or loop diuretic

Exclusion Criteria:

* Has known history of secondary hypertension
* Has symptomatic orthostatic hypotension
* Has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3×upper limit of normal (ULN)
* Has total serum bilirubin >1.5×ULN
* Has international normalized ratio (INR) >1.5
* Has serum potassium >4.8 mEq/L
* Has estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m^2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11000 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2030-10-29 (Estimated); Study Completion 2030-10-29 (Estimated)

PRIMARY OUTCOMES:
Time to First Occurrence of a Composite Endpoint of Cardiovascular (CV) Death, Nonfatal Myocardial Infarction (MI), Nonfatal Stroke, or Heart Failure (HF) Event (Hospitalization for HF or Urgent HF Visit) | Up to approximately 5 years

SECONDARY OUTCOMES:
Change from Baseline in Mean Seated Office Systolic Blood Pressure (SBP) at Month 6 | Baseline and Month 6
Time to First Occurrence of a Composite Endpoint of CV Death, Nonfatal MI, or Nonfatal Stroke | Up to approximately 5 years
Composite Endpoint of CV Death and Total (First and Subsequent) HF Events (Hospitalization for HF or Urgent HF Visit) | Up to approximately 5 years
Time to First Occurrence of Composite Endpoint of CV death, Nonfatal MI, Nonfatal Stroke, or Coronary Revascularization | Up to approximately 5 years
Time to All-cause Death | Up to approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals Inc
Locations (29):
- United States (29):
  - Clinical Trial Site, Phoenix, Arizona
  - Clinical Trial Site, Tucson, Arizona
  - Clinical Trial Site, Little Rock, Arkansas
  - Clinical Trial Site, Escondido, California
  - Clinical Trial Site, Brandon, Florida
  - Clinical Trial Site, Jacksonville, Florida
  - Clinical Trial Site, Melbourne, Florida
  - Clinical Trial Site, Miami, Florida
  - Clinical Trial Site, Orlando, Florida
  - Clinical Trial Site, Palm Springs, Florida
  - Clinical Trial Site, Tampa, Florida
  - Clinical Trial Site, Flossmoor, Illinois
  - Clinical Trial Site, Evansville, Indiana
  - Clinical Trial Site, Valparaiso, Indiana
  - Clinical Trial Site, Albuquerque, New Mexico
  - Clinical Trial Site, New Windsor, New York
  - Clinical Trial Site, Fargo, North Dakota
  - Clinical Trial Site, Cincinnati, Ohio
  - Clinical Trial Site, Columbus, Ohio
  - Clinical Trial Site, Maumee, Ohio
  - Clinical Trial Site, Chattanooga, Tennessee
  - Clinical Trial Site, Knoxville, Tennessee
  - Clinical Trial Site, Houston, Texas
  - Clinical Trial Site, McKinney, Texas
  - Clinical Trial Site, Mesquite, Texas
  - Clinical Trial Site, Missouri City, Texas
  - Clinical Trial Site, Plano, Texas
  - Clinical Trial Site, Richmond, Texas
  - Clinical Trial Site, Bountiful, Utah

IPD SHARING:
Plan to Share IPD: Yes
Phase 2-4 trials:
  Access to anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the US and/or the EU.
  Access to data may be declined where there is likelihood a patient could be identified or other feasibility issue, where there is a potential conflict of interest, a planned business activities or an actual or potential competitive risk. Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Timeframes for data access may vary and can take up to 6 months or more.
  Requests for access to data can be submitted via the website www.vivli.org. Questions can also be directed to datasharing@alnylam.com.